CLINICAL TRIAL: NCT00484120
Title: Proof-of Concept Study to Evaluate the Safety and Analgesic Efficacy of Topical 3%-Diclofenac-Nano-Emulsion Cream Versus Placebo for Knee Osteoarthritis
Brief Title: Proof-of Concept Study of Topical 3%-Diclofenac-Nano-Emulsion Cream for Knee OA Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmos (Industry)
Responsible Party: Clinical Team, Pharmos Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PH-2007-2
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-08

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Diclofenac; Nano-emulsion
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 3% Diclofenac NE cream
  Interventions: Drug: 3%-Diclofenac-Nano-Emulsion Cream
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: 3%-Diclofenac-Nano-Emulsion Cream — 3%-Diclofenac-Nano-Emulsion Cream
  Arms: 1
Drug: Placebo cream — Placebo cream
  Arms: 2

SUMMARY:
This study valuates the safety and efficacy of treatment with 3% Diclofenac Nano-Emulsion Cream versus Placebo in subjects with osteoarthritis of the knee.

DETAILED DESCRIPTION:
This will be a multi-center, double-blind, placebo-controlled, multiple-dose, parallel treatment study. A total of 126 subjects will be randomized to receive either 3%-Diclofenac-NE cream or a placebo cream respectively. Following screening and a washout period from previous treatments subjects will be enrolled and will self-apply the study medication. During the study, subjects will apply 3%-Diclofenac-NE or placebo cream three times daily for 28 days and complete a home-diary. Subjects will visit the clinic at mid-treatment for a follow up examination and again for a final examination at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 50 years of age and above.
2. Patients with primary osteoarthritis in at least a single knee joint, grade 2 or 3 based on the Kellgren and Lawrence classification system.
3. Radiographic evidence consistent with OA carried out within the 6 months before screening.
4. Pain should have been present for at least half of the days in the previous month and for at least 48h prior to the screening visit.
5. Eligible subjects must have used an oral, topical or rectal NSAID within the past 6 months before screening.
6. At baseline, after a 1 week withdrawal period of analgesic/anti-inflammatory medications, subjects should have a flare of pain.
7. Able to read, comprehend, and sign the consent form.
8. Examined by the authorized physician and medically cleared to participate in the study.
9. In general good health and have no contraindications to any of the investigational medicinal products.

Exclusion Criteria:

1. Secondary osteoarthritis.
2. Presence of a serious or unstable medical condition (e.g., malignancy, severe neurological impairment or uncontrolled hypertension) or poor general health interfering with compliance or assessment at the study physician's discretion.
3. OA causing significant pain in any joint other than the knees.
4. Any other rheumatic or non-rheumatic joint disease or any other painful condition within the past month (e.g. fibromyalgia).
5. Knee surgery or other knee trauma at any time during the previous year or subjects for whom a treatment is planned within the study period that could alter the degree or nature of pain (e.g. arthroscopic techniques, osteotomy, joint replacement surgery etc.).
6. Active or history of gastrointestinal ulceration or bleeding within the past 5 years.
7. Presence of a significant active psychiatric disorder including major depression or subjects receiving anti-psychotic medication.
8. Existence of any dermatological condition on the knee.
9. Subjects with disabling congestive heart failure (CHF), angina, pulmonary disease.
10. Clinically significant abnormal blood results.
11. Subjects cannot have had an arthrocentesis prior or during the study.
12. Concomitant treatment with physical and/or occupational therapy.
13. Prior use of any type of NSAID or other analgesic before taking the first dose of investigational medicinal product. Rescue treatment will be allowed during the study
14. Change in sedative or CNS/psychotropic agent within the past month.
15. Chronic treatment with anticoagulants (e.g. Warfarin).
16. Subjects under treatment with corticosteroids.
17. Subjects using topical analgesics including OTC products.
18. Females who are pregnant, lactating, of child-bearing potential, or post-menopausal for less than 2 years and not using a medically approved method of contraception (i.e., oral, transdermal, or implanted contraceptives, intrauterine device, diaphragm, condom, abstinence, or surgical sterility), or females who test positive on a urine-based pregnancy test.
19. Active alcoholism or substance abuse.
20. Has taken an investigational drug or has used an investigational device within the past 30 days.
21. History of hypersensitivity and/or idiosyncrasy to diclofenac or excipients employed in this study, aspirin or other NSAIDS.
22. Has previously been entered into this study.
23. Any condition that in the investigator's judgement precludes participation in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2007-06; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Analgesic activity as measured by the WOMAC pain subscale. | 1 month

SECONDARY OUTCOMES:
Patient's daily pain assessment in the home diary. | 1 month
Pain on walking. | 1 month
Safety and Tolerability. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Eisenberg Elon, MD, Principal Investigator — Rambam Health Care Campus
Locations (4):
- Israel (4):
  - Barzilai Medical Center, Ashkelon, Israel
  - Rabin Medical Center, Petah Tikva, Israel
  - Rambam Medical Center, Haifa
  - Sourasky Medical Center, Tel Aviv